CLINICAL TRIAL: NCT03611803
Title: EFFECTS OF ROBOTIC-ASSISTED GAIT TRAINING ON THE VASCULAR HEALTH OF INDIVIDUALS WITH SPINAL CORD INJURY
Brief Title: EFFECTS OF ROBOTIC TRAINING ON VASCULAR HEALTH OF INDIVIDUALS WITH SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Hobbs Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Faulkner_Ekso_SCI
Record Dates: First submitted 2018-06-28; First posted 2018-08-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Exercise; Spinal Cord Injuries
Keywords: Robotic-assisted gait training; SCI; Ambulatory activity
MeSH Terms: conditions — Motor Activity; Spinal Cord Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ekso Group (Experimental)
  Interventions: Device: Physiotherapy + Robotic-device
- Control (Active Comparator)
  Interventions: Other: Physiotherapy only

INTERVENTIONS:
Device: Physiotherapy + Robotic-device — Daily use of an exoskeleton (robotic-device) on 5 successive days as well as daily physiotherapy sessions
  Arms: Ekso Group
Other: Physiotherapy only — Participants will engage in daily physiotherapy sessions (without the exoskeleton) and/or home-based sit-to-stand exercises
  Arms: Control

SUMMARY:
Robotic devices may be used to help the gait and balance of individuals with Spinal Cord Injury (SCI). However, as such devices may allow individuals to engage in physical activity in an upright position, there may be significant benefit on the vascular health of patients with SCI. This study will assess the effect of a robotic-assisted gait-training (exoskeleton) program on central and peripheral hemodynamic markers in people with SCI.

DETAILED DESCRIPTION:
Individuals with spinal cord injury (SCI) have an accelerated trajectory of aging in the cardiovascular system compared with same-age individuals in the general population,and accordingly, have a higher rate of cardiovascular mortality. For example, SCI is significantly associated with an increased risk of heart disease (odds ratio = 2.72) and stroke (odds ratio = 3.72).This is at least partially attributed to their impaired blood pressure regulation as a consequence of the autonomic nervous system dysfunction, physical inactivity and increased sedentary time. As such, there is a pressing need to identify practical strategies for increasing physical activity and decreasing sedentary time.

Robotic-assisted gait training (RGT) is used in the rehabilitation of patients with SCI, although individual access is often limited and infrequent. Task-specific stepping practice enhances the afferent feedback associated with normal locomotion and can induce plasticity in the involved motor centers. As RGT enables practitioners to increase the intensity and total duration of physical activity whilst maintaining a physiological gait pattern, there may be significant benefit for people with SCI to manage their risk of cardiovascular disease (CVD). This may be evident if an individual with SCI has regular and continued access to such technology. However, there is a paucity of research which has considered the vascular benefit of implementing robotic-assisted training for people with SCI as most research focuses on outcome measures such as gait velocity, gait distance, leg strength, balance and spasticity.Further, while this technology may be practical in terms of application, the cost is currently prohibitive. Thus, prior to advocating resource intensive longitudinal randomized control trials, there's a need for short-term trials using established measures of cardiovascular health.

The purpose of this study is to assess the effect of a RGT (exoskeleton) program on central and peripheral hemodynamic markers in people with SCI.

ELIGIBILITY:
Inclusion Criteria:

* SCI diagnosis
* Meet the manufacturer's guidelines with regards to weight (< 100 kg) and height (between 1.57 m and 1.93 m).
* Standing at least three times a week with therapist support
* SCI classified according to the American Spinal Injury Association (ASIA) scale, as either ASIA A (Complete SCI), ASIA B (Sensory incomplete SCI), ASIA C (Motor incomplete SCI)

Exclusion Criteria:

* Restricted range of motion in their lower limbs
* Uncontrolled high levels of muscle spasticity
* Significant problems managing their blood pressure,
* Any concerns with their bone density (e.g., osteoporosis, etc.).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Augmentation index | Assessed at Baseline and Through study completion (1 week after baseline).
  Measured on the left, upper arm, in duplicate and following a 20 minute supine rest using a SphygmoCor XCEL.

SECONDARY OUTCOMES:
Change in Central Blood pressure | Assessed at Baseline and Through study completion (1 week after baseline).
  Measured on the left, upper arm, in duplicate and following a 20 minute supine rest using a SphygmoCor XCEL.
Change in Peripheral blood pressure | Assessed at Baseline and Through study completion (1 week after baseline).
  Measured on the left, upper arm, in duplicate and following a 20 minute supine rest using a SphygmoCor XCEL.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sport, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faulkner J, Martinelli L, Cook K, Stoner L, Ryan-Stewart H, Paine E, Hobbs H, Lambrick D. Effects of robotic-assisted gait training on the central vascular health of individuals with spinal cord injury: A pilot study. J Spinal Cord Med. 2021 Mar;44(2):299-305. doi: 10.1080/10790268.2019.1656849. Epub 2019 Sep 16. PMID 31525137